CLINICAL TRIAL: NCT04790708
Title: Peptide Receptor Radionuclide Therapy (PRRT) in Tumors With High Expression of Somatostatin Receptors
Brief Title: Peptide Receptor Radionuclide Therapy (PRRT) in Tumors With High Expression of Somatostatin Receptors (Phase 2)
Acronym: FENET-2016
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital of Ferrara (Other)
Responsible Party: Principal Investigator, Mirco Bartolomei, MD, Director of Nuclear Medicine Unit, University Hospital of Ferrara
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 160990; 2016-005129-35 (EudraCT Number)
Record Dates: First submitted 2021-03-02; First posted 2021-03-10 (Actual); Last update posted 2021-03-10 (Actual); Status verified 2021-03

CONDITIONS: Neuroendocrine Tumors; Peptide Receptor Radionuclide Therapy (PRRT)
Keywords: Neuroendocrine Tumors; 90Y; 177Lu; PRRT
MeSH Terms: conditions — Neuroendocrine Tumors | interventions — Lutetium-177; 177Lu-octreotide, DOTA(0)-Tyr(3)-; Yttrium-90; 90Y-octreotide, DOTA-Tyr(3)-

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- Midgut NETs (Experimental): 75 patients affected by non-functional and functional NETs arising from: stomach, duodenum, jejunum, ileum, colon and rectum.
  Interventions: Radiation: Lutetium-177 (177Lu)-DOTATOC; Radiation: Yttrium-90 (90Y)-DOTATOC; Radiation: 177Lu-DOTATOC + 90Y-DOTATOC; Radiation: Re-treatment 177Lu-DOTATOC; Radiation: Re-treatment 90Y-DOTATOC
- Pancreatic NETs (Experimental): 75 patients affected by non-functional and functional NETs arising from Pancreas.
  Interventions: Radiation: Lutetium-177 (177Lu)-DOTATOC; Radiation: Yttrium-90 (90Y)-DOTATOC; Radiation: 177Lu-DOTATOC + 90Y-DOTATOC; Radiation: Re-treatment 177Lu-DOTATOC; Radiation: Re-treatment 90Y-DOTATOC
- Bronchial NETs (Experimental): 25 patients affected by non-functional and functional Bronchial NETs.
  Interventions: Radiation: Lutetium-177 (177Lu)-DOTATOC; Radiation: Yttrium-90 (90Y)-DOTATOC; Radiation: 177Lu-DOTATOC + 90Y-DOTATOC; Radiation: Re-treatment 177Lu-DOTATOC; Radiation: Re-treatment 90Y-DOTATOC
- Sympathetic-Adrenergic axis NEts (Experimental): 25 patients affected by non-functional and functional: Pheochromocytoma, Paraganglioma and Neuroblastoma
  Interventions: Radiation: Lutetium-177 (177Lu)-DOTATOC; Radiation: Yttrium-90 (90Y)-DOTATOC; Radiation: 177Lu-DOTATOC + 90Y-DOTATOC; Radiation: Re-treatment 177Lu-DOTATOC; Radiation: Re-treatment 90Y-DOTATOC
- Other Nets (Experimental): 25 patients affected by non-functional and functional NETs arising from Skin, Thyroid (medullary thyroid and anaplastic cancer) and Parathyroids.
  Interventions: Radiation: Lutetium-177 (177Lu)-DOTATOC; Radiation: Yttrium-90 (90Y)-DOTATOC; Radiation: 177Lu-DOTATOC + 90Y-DOTATOC; Radiation: Re-treatment 177Lu-DOTATOC; Radiation: Re-treatment 90Y-DOTATOC
- Cancers of Unknown Primary Origin (CUP) NETs (Experimental): 25 patients affected by non-functional and functional unknown primary NETs
  Interventions: Radiation: Lutetium-177 (177Lu)-DOTATOC; Radiation: Yttrium-90 (90Y)-DOTATOC; Radiation: 177Lu-DOTATOC + 90Y-DOTATOC; Radiation: Re-treatment 177Lu-DOTATOC; Radiation: Re-treatment 90Y-DOTATOC

INTERVENTIONS:
Radiation: Lutetium-177 (177Lu)-DOTATOC — 5 cycles of 3,7 e 5,55 gigabequerel (GBq) of 177Lu-DOTATOC every 8-10 weeks. Cumulative activity: 18,5 e 27,75 GBq
  Other Names: "MONO"
Radiation: Yttrium-90 (90Y)-DOTATOC — 5 cycles of 1,85 e 2,775 GBq of 90Y-DOTATOC every 8-10 weeks. Cumulative activity: 9,25 e 13,875 GBq
Radiation: 177Lu-DOTATOC + 90Y-DOTATOC — 3 cycles of 3,7 e 5,55 GBq of 177Lu-DOTATOC alternated with 2 cycles of 1,85 e 2,775 GBq of 90Y-DOTATOC every 8-10 weeks.
  Cumulative activity: 18,5 e 27,75 GBq of 177Lu-DOTATOC and 9,25 e 13,875 GBq of 90Y-DOTATOC
  Other Names: "DUO"
Radiation: Re-treatment 177Lu-DOTATOC — 3 cycles of 3,7 e 5,55 GBq of 177Lu-DOTATOC every 8-10weeks. Cumulative activity: 11,1 e 16,65 GBq of 177Lu-DOTATOC
Radiation: Re-treatment 90Y-DOTATOC — 3 cycles of 1,85 e 2,775 GBq of 90Y-DOTATOC every 8-10 weeks Cumulative activity: 5,55 e 8,325 GBq of 90Y-DOTATOC

SUMMARY:
The rationale behind the purpose of this study lays on:

* the evidence that PRRT could represent a valuable treatment for the majority of patients with neuroendocrine tumor (NET) in disease progression, operated or inoperable, presenting lesions expressing somatostatin receptors and for which standard treatments are not already available;
* the current impossibility of acquiring on the market radiolabelled analogues of somatostatin used for PRRT with marketing authorisation;
* the need to collect a larger case history than in previous studies;
* the need to stratify the various histotypes based on the response obtained;
* the need to define new treatment schemes that guarantee the maximum efficacy and the lowest possible toxicity - with low cumulative (and per cycle) activities radiopharmaceutical and according to the concept of dose hyperfractionation - with a view to an optimal balance between risk and benefit.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age ≥18 years, of both sexes, of any ethnicity;
* 2. Cyto-histological and immunohistochemical diagnosis of NET;
* 3. Evaluation of the cell proliferation index by studying Ki-67 and / or E3 ubiquitin-protein ligase (MIB-1).
* 4. Illness measurable according to RECIST 1.1 criteria by imaging conventional (CT with contrast medium or MRI with contrast medium) not earlier than two months with respect to enrollment;
* 5. Elevated expression of somatostatin receptors documented by PET-CT with 68Ga-DOTATOC in the target lesion (s). It is defined as "high expression of somatostatin receptors "a ratio of Maximum standardized uptake value (SUVmax) lesion / Mean standardized uptake value (SUVmean) muscle ≥ 4: 1 calculated with semi-quantitative analysis on examination PET-CT with 68Ga-DOTATOC;
* 6. Dosage of Chromogranin A (and any other specific markers) not prior to two months of enrollment;
* 7. Evaluation of glucose metabolism in the target lesion (s) by PET-CT with 18F-FDG;
* 8. Preserved haematological, hepatic and renal parameters, in particular: white blood cells ≥2500 / μL; platelets ≥ 90000 / μL; hemoglobin ≥ 9 gr / dL; creatinine ≤ 2 mg / dL; bilirubin ≤ 2.5 mg / dL
* 9. Eastern Cooperative Oncology Group (ECOG) performance status ≤2;
* 10. Life expectancy ≥ 6 months;
* 11. Stable or progressive disease, at any stage, both in operated patients that inoperable;
* 12. Absence of standard treatments already documented and of equal effectiveness;
* 13. Absence of surgical, chemotherapy and / or radiotherapy treatments for at least 30 days. On the other hand, patients in therapy with somatostatin analogues or biologics, such as mechanistic target of rapamycin (m-TOR) inhibitors;
* 14. Voluntary participation in the study by signing the consent form informed, after reading and complete understanding of the information notes.

Exclusion Criteria:

* 1. Lack of the requirements listed above;
* 2. State of pregnancy;
* 3. Breastfeeding and relative refusal to suspend breastfeeding;
* 4. Participation in another therapeutic experimental clinical protocol in the four weeks prior to the PRRT;
* 5. Bone marrow invasion of disease> 25% confirmed;
* 6. Previous extensive radiotherapy treatments.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2018-07-02 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Disease Control Rate | 12 months
  Post-treatment evaluation will be performed with:
  * a clinical examination;
  * a comparative morphological re-evaluation, using version 1.1 of Response evaluation criteria in solid tumors (RECIST criteria) on Computed Tomography (CT);
  * a comparative functional re-evaluation, performed both on 18F-2-fluoro-2-deoxy-D-glucose (18F-FDG) positron emission computed tomography (PET/CT) and Gallium-68 (68Ga)-DOTATOC PET/CT using visual and semi-quantitative parameters (such as SUVmax).
  Based on all these parameters, Disease Control Rate will be labelled as: Complete Response (CR), Partial Response (PR), Stable Disease (SD), or Progression Disease (PD).

SECONDARY OUTCOMES:
Progression Free Survival | 6 months
  Progression free survival is defined as the time intercurrent from treatment start to the date of first observation of documented disease progression or death due to any cause.
Overall Survival | 6 months
  Overall survival is defined as the time intercurrent from treatment start to the date of death due to any cause, or the date of last contact.
Evaluation of PRRT Safety | 6 months
  The evaluation of Treatment-Emergent Adverse Events, defined as any G3/G4 toxicity. The evaluation will be performed during every treatment cycle and after 12, 18, 24, 30, 36 and 42 months after the last treatment cycle and will be based on version 4.0 of Common Terminology Criteria for Adverse Events (CTC-AE) toxicity criteria.
Evaluation of Quality of Life | 6 months
  Quality of Life (QoL) will be evaluated with quality of life questionnaire, version 3 (QLQ-C30) by European Organisation for Research and Treatment of Cancer (EORTC). The questionnaire includes five functional scales, three symptom scales, a global health status / QoL scale, and six single items.
  All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Ferrara, Ferrara, Italy

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Smit Duijzentkunst DA, Kwekkeboom DJ, Bodei L. Somatostatin Receptor 2-Targeting Compounds. J Nucl Med. 2017 Sep;58(Suppl 2):54S-60S. doi: 10.2967/jnumed.117.191015. PMID 28864613
- [Background] Modlin IM, Lye KD, Kidd M. A 5-decade analysis of 13,715 carcinoid tumors. Cancer. 2003 Feb 15;97(4):934-59. doi: 10.1002/cncr.11105. PMID 12569593
- [Background] Teunissen JJ, Kwekkeboom DJ, Valkema R, Krenning EP. Nuclear medicine techniques for the imaging and treatment of neuroendocrine tumours. Endocr Relat Cancer. 2011 Oct 17;18 Suppl 1:S27-51. doi: 10.1530/ERC-10-0282. Print 2011 Oct. PMID 22005114
- [Background] Yao JC, Hassan M, Phan A, Dagohoy C, Leary C, Mares JE, Abdalla EK, Fleming JB, Vauthey JN, Rashid A, Evans DB. One hundred years after "carcinoid": epidemiology of and prognostic factors for neuroendocrine tumors in 35,825 cases in the United States. J Clin Oncol. 2008 Jun 20;26(18):3063-72. doi: 10.1200/JCO.2007.15.4377. PMID 18565894
- [Background] Hemminki K, Li X. Incidence trends and risk factors of carcinoid tumors: a nationwide epidemiologic study from Sweden. Cancer. 2001 Oct 15;92(8):2204-10. doi: 10.1002/1097-0142(20011015)92:83.0.co;2-r. PMID 11596039
- [Background] Modlin IM, Oberg K, Chung DC, Jensen RT, de Herder WW, Thakker RV, Caplin M, Delle Fave G, Kaltsas GA, Krenning EP, Moss SF, Nilsson O, Rindi G, Salazar R, Ruszniewski P, Sundin A. Gastroenteropancreatic neuroendocrine tumours. Lancet Oncol. 2008 Jan;9(1):61-72. doi: 10.1016/S1470-2045(07)70410-2. PMID 18177818
- [Background] Kloppel G, Couvelard A, Perren A, Komminoth P, McNicol AM, Nilsson O, Scarpa A, Scoazec JY, Wiedenmann B, Papotti M, Rindi G, Plockinger U; Mallorca Consensus Conference participants; European Neuroendocrine Tumor Society. ENETS Consensus Guidelines for the Standards of Care in Neuroendocrine Tumors: towards a standardized approach to the diagnosis of gastroenteropancreatic neuroendocrine tumors and their prognostic stratification. Neuroendocrinology. 2009;90(2):162-6. doi: 10.1159/000182196. Epub 2009 Aug 28. No abstract available. PMID 19060454
- [Background] Rindi G, Kloppel G, Couvelard A, Komminoth P, Korner M, Lopes JM, McNicol AM, Nilsson O, Perren A, Scarpa A, Scoazec JY, Wiedenmann B. TNM staging of midgut and hindgut (neuro) endocrine tumors: a consensus proposal including a grading system. Virchows Arch. 2007 Oct;451(4):757-62. doi: 10.1007/s00428-007-0452-1. Epub 2007 Aug 3. PMID 17674042
- [Background] Scoazec JY, Couvelard A; pour le reseau TENpath (reseau national d'expertise pour le diagnostic anatomopathologique des tumeurs neuroendocrines malignes de l'adulte, sporadiques et familiales). [The new WHO classification of digestive neuroendocrine tumors]. Ann Pathol. 2011 Apr;31(2):88-92. doi: 10.1016/j.annpat.2011.01.001. Epub 2011 Mar 26. French. PMID 21601112
- [Background] Volante M, Gatti G, Papotti M. Classification of lung neuroendocrine tumors: lights and shadows. Endocrine. 2015 Nov;50(2):315-9. doi: 10.1007/s12020-015-0578-x. Epub 2015 Mar 21. PMID 25795289
- [Background] Warner RR. Enteroendocrine tumors other than carcinoid: a review of clinically significant advances. Gastroenterology. 2005 May;128(6):1668-84. doi: 10.1053/j.gastro.2005.03.078. PMID 15887158
- [Background] Massironi S, Sciola V, Peracchi M, Ciafardini C, Spampatti MP, Conte D. Neuroendocrine tumors of the gastro-entero-pancreatic system. World J Gastroenterol. 2008 Sep 21;14(35):5377-84. doi: 10.3748/wjg.14.5377. PMID 18803349
- [Background] Ramage JK, Davies AH, Ardill J, Bax N, Caplin M, Grossman A, Hawkins R, McNicol AM, Reed N, Sutton R, Thakker R, Aylwin S, Breen D, Britton K, Buchanan K, Corrie P, Gillams A, Lewington V, McCance D, Meeran K, Watkinson A; UKNETwork for Neuroendocrine Tumours. Guidelines for the management of gastroenteropancreatic neuroendocrine (including carcinoid) tumours. Gut. 2005 Jun;54 Suppl 4(Suppl 4):iv1-16. doi: 10.1136/gut.2004.053314. No abstract available. PMID 15888809
- [Background] de Baere T, Deschamps F, Tselikas L, Ducreux M, Planchard D, Pearson E, Berdelou A, Leboulleux S, Elias D, Baudin E. GEP-NETS update: Interventional radiology: role in the treatment of liver metastases from GEP-NETs. Eur J Endocrinol. 2015 Apr;172(4):R151-66. doi: 10.1530/EJE-14-0630. Epub 2014 Nov 10. PMID 25385817
- [Background] Jann H, Denecke T, Koch M, Pape UF, Wiedenmann B, Pavel M. Impact of octreotide long-acting release on tumour growth control as a first-line treatment in neuroendocrine tumours of pancreatic origin. Neuroendocrinology. 2013;98(2):137-43. doi: 10.1159/000353785. Epub 2013 Aug 13. PMID 23797176
- [Background] Bison SM, Konijnenberg MW, Melis M, Pool SE, Bernsen MR, Teunissen JJ, Kwekkeboom DJ, de Jong M. Peptide receptor radionuclide therapy using radiolabeled somatostatin analogs: focus on future developments. Clin Transl Imaging. 2014;2(1):55-66. doi: 10.1007/s40336-014-0054-2. Epub 2014 Mar 5. PMID 24765618
- [Background] Rajekar H, Bogammana K, Stubbs RS. Selective internal radiation therapy for gastrointestinal neuroendocrine tumour liver metastases: a new and effective modality for treatment. Int J Hepatol. 2011;2011:404916. doi: 10.4061/2011/404916. Epub 2011 Nov 15. PMID 22164335
- [Background] Panzuto F, Rinzivillo M, Fazio N, de Braud F, Luppi G, Zatelli MC, Lugli F, Tomassetti P, Riccardi F, Nuzzo C, Brizzi MP, Faggiano A, Zaniboni A, Nobili E, Pastorelli D, Cascinu S, Merlano M, Chiara S, Antonuzzo L, Funaioli C, Spada F, Pusceddu S, Fontana A, Ambrosio MR, Cassano A, Campana D, Carteni G, Appetecchia M, Berruti A, Colao A, Falconi M, Delle Fave G. Real-world study of everolimus in advanced progressive neuroendocrine tumors. Oncologist. 2015 May;20(5):570. doi: 10.1634/theoncologist.2014-0037erratum. No abstract available. PMID 25956900
- [Background] Dong M, Phan AT, Yao JC. New strategies for advanced neuroendocrine tumors in the era of targeted therapy. Clin Cancer Res. 2012 Apr 1;18(7):1830-6. doi: 10.1158/1078-0432.CCR-11-2105. Epub 2012 Feb 15. PMID 22338018
- [Background] Kulke MH, Bendell J, Kvols L, Picus J, Pommier R, Yao J. Evolving diagnostic and treatment strategies for pancreatic neuroendocrine tumors. J Hematol Oncol. 2011 Jun 14;4:29. doi: 10.1186/1756-8722-4-29. PMID 21672194
- [Background] Bodei L, Mueller-Brand J, Baum RP, Pavel ME, Horsch D, O'Dorisio MS, O'Dorisio TM, Howe JR, Cremonesi M, Kwekkeboom DJ, Zaknun JJ. The joint IAEA, EANM, and SNMMI practical guidance on peptide receptor radionuclide therapy (PRRNT) in neuroendocrine tumours. Eur J Nucl Med Mol Imaging. 2013 May;40(5):800-16. doi: 10.1007/s00259-012-2330-6. PMID 23389427
- [Background] Reubi JC, Schaer JC, Laissue JA, Waser B. Somatostatin receptors and their subtypes in human tumors and in peritumoral vessels. Metabolism. 1996 Aug;45(8 Suppl 1):39-41. doi: 10.1016/s0026-0495(96)90077-3. PMID 8769377
- [Background] Kwekkeboom DJ, Krenning EP. Somatostatin receptor imaging. Semin Nucl Med. 2002 Apr;32(2):84-91. doi: 10.1053/snuc.2002.31022. PMID 11965603
- [Background] Reubi JC, Waser B, Schaer JC, Laissue JA. Somatostatin receptor sst1-sst5 expression in normal and neoplastic human tissues using receptor autoradiography with subtype-selective ligands. Eur J Nucl Med. 2001 Jul;28(7):836-46. doi: 10.1007/s002590100541. PMID 11504080
- [Background] Reubi JC, Schar JC, Waser B, Wenger S, Heppeler A, Schmitt JS, Macke HR. Affinity profiles for human somatostatin receptor subtypes SST1-SST5 of somatostatin radiotracers selected for scintigraphic and radiotherapeutic use. Eur J Nucl Med. 2000 Mar;27(3):273-82. doi: 10.1007/s002590050034. PMID 10774879
- [Background] Ducreux M, Ruszniewski P, Chayvialle JA, Blumberg J, Cloarec D, Michel H, Raymond JM, Dupas JL, Gouerou H, Jian R, Genestin E, Hammel P, Rougier P. The antitumoral effect of the long-acting somatostatin analog lanreotide in neuroendocrine tumors. Am J Gastroenterol. 2000 Nov;95(11):3276-81. doi: 10.1111/j.1572-0241.2000.03210.x. PMID 11095353
- [Background] Rinke A, Muller HH, Schade-Brittinger C, Klose KJ, Barth P, Wied M, Mayer C, Aminossadati B, Pape UF, Blaker M, Harder J, Arnold C, Gress T, Arnold R; PROMID Study Group. Placebo-controlled, double-blind, prospective, randomized study on the effect of octreotide LAR in the control of tumor growth in patients with metastatic neuroendocrine midgut tumors: a report from the PROMID Study Group. J Clin Oncol. 2009 Oct 1;27(28):4656-63. doi: 10.1200/JCO.2009.22.8510. Epub 2009 Aug 24. PMID 19704057
- [Background] Caplin ME, Pavel M, Cwikla JB, Phan AT, Raderer M, Sedlackova E, Cadiot G, Wolin EM, Capdevila J, Wall L, Rindi G, Langley A, Martinez S, Blumberg J, Ruszniewski P; CLARINET Investigators. Lanreotide in metastatic enteropancreatic neuroendocrine tumors. N Engl J Med. 2014 Jul 17;371(3):224-33. doi: 10.1056/NEJMoa1316158. PMID 25014687
- [Background] Krenning EP, Kwekkeboom DJ, Bakker WH, Breeman WA, Kooij PP, Oei HY, van Hagen M, Postema PT, de Jong M, Reubi JC, et al. Somatostatin receptor scintigraphy with [111In-DTPA-D-Phe1]- and [123I-Tyr3]-octreotide: the Rotterdam experience with more than 1000 patients. Eur J Nucl Med. 1993 Aug;20(8):716-31. doi: 10.1007/BF00181765. PMID 8404961
- [Background] Reubi JC. Somatostatin and other Peptide receptors as tools for tumor diagnosis and treatment. Neuroendocrinology. 2004;80 Suppl 1:51-6. doi: 10.1159/000080742. PMID 15477718
- [Background] Bombardieri E, Seregni E, Villano C, Chiti A, Bajetta E. Position of nuclear medicine techniques in the diagnostic work-up of neuroendocrine tumors. Q J Nucl Med Mol Imaging. 2004 Jun;48(2):150-63. PMID 15243410
- [Background] Lebtahi R, Cadiot G, Sarda L, Daou D, Faraggi M, Petegnief Y, Mignon M, le Guludec D. Clinical impact of somatostatin receptor scintigraphy in the management of patients with neuroendocrine gastroenteropancreatic tumors. J Nucl Med. 1997 Jun;38(6):853-8. PMID 9189129
- [Background] Chiti A, Fanti S, Savelli G, Romeo A, Bellanova B, Rodari M, van Graafeiland BJ, Monetti N, Bombardieri E. Comparison of somatostatin receptor imaging, computed tomography and ultrasound in the clinical management of neuroendocrine gastro-entero-pancreatic tumours. Eur J Nucl Med. 1998 Oct;25(10):1396-403. doi: 10.1007/s002590050314. PMID 9818279
- [Background] Chiti A, Briganti V, Fanti S, Monetti N, Masi R, Bombardieri E. Results and potential of somatostatin receptor imaging in gastroenteropancreatic tract tumours. Q J Nucl Med. 2000 Mar;44(1):42-9. PMID 10932600
- [Background] Kowalski J, Henze M, Schuhmacher J, Macke HR, Hofmann M, Haberkorn U. Evaluation of positron emission tomography imaging using [68Ga]-DOTA-D Phe(1)-Tyr(3)-Octreotide in comparison to [111In]-DTPAOC SPECT. First results in patients with neuroendocrine tumors. Mol Imaging Biol. 2003 Jan-Feb;5(1):42-8. doi: 10.1016/s1536-1632(03)00038-6. PMID 14499161
- [Background] Buchmann I, Henze M, Engelbrecht S, Eisenhut M, Runz A, Schafer M, Schilling T, Haufe S, Herrmann T, Haberkorn U. Comparison of 68Ga-DOTATOC PET and 111In-DTPAOC (Octreoscan) SPECT in patients with neuroendocrine tumours. Eur J Nucl Med Mol Imaging. 2007 Oct;34(10):1617-26. doi: 10.1007/s00259-007-0450-1. Epub 2007 May 23. PMID 17520251
- [Background] Hofmann M, Maecke H, Borner R, Weckesser E, Schoffski P, Oei L, Schumacher J, Henze M, Heppeler A, Meyer J, Knapp H. Biokinetics and imaging with the somatostatin receptor PET radioligand (68)Ga-DOTATOC: preliminary data. Eur J Nucl Med. 2001 Dec;28(12):1751-7. doi: 10.1007/s002590100639. Epub 2001 Oct 31. PMID 11734911
- [Background] Wild D, Schmitt JS, Ginj M, Macke HR, Bernard BF, Krenning E, De Jong M, Wenger S, Reubi JC. DOTA-NOC, a high-affinity ligand of somatostatin receptor subtypes 2, 3 and 5 for labelling with various radiometals. Eur J Nucl Med Mol Imaging. 2003 Oct;30(10):1338-47. doi: 10.1007/s00259-003-1255-5. Epub 2003 Aug 21. PMID 12937948
- [Background] Ambrosini V, Campana D, Bodei L, Nanni C, Castellucci P, Allegri V, Montini GC, Tomassetti P, Paganelli G, Fanti S. 68Ga-DOTANOC PET/CT clinical impact in patients with neuroendocrine tumors. J Nucl Med. 2010 May;51(5):669-73. doi: 10.2967/jnumed.109.071712. Epub 2010 Apr 15. PMID 20395323
- [Background] Antunes P, Ginj M, Zhang H, Waser B, Baum RP, Reubi JC, Maecke H. Are radiogallium-labelled DOTA-conjugated somatostatin analogues superior to those labelled with other radiometals? Eur J Nucl Med Mol Imaging. 2007 Jul;34(7):982-93. doi: 10.1007/s00259-006-0317-x. Epub 2007 Jan 16. PMID 17225119
- [Background] Gabriel M, Decristoforo C, Kendler D, Dobrozemsky G, Heute D, Uprimny C, Kovacs P, Von Guggenberg E, Bale R, Virgolini IJ. 68Ga-DOTA-Tyr3-octreotide PET in neuroendocrine tumors: comparison with somatostatin receptor scintigraphy and CT. J Nucl Med. 2007 Apr;48(4):508-18. doi: 10.2967/jnumed.106.035667. PMID 17401086
- [Background] Hofman MS, Kong G, Neels OC, Eu P, Hong E, Hicks RJ. High management impact of Ga-68 DOTATATE (GaTate) PET/CT for imaging neuroendocrine and other somatostatin expressing tumours. J Med Imaging Radiat Oncol. 2012 Feb;56(1):40-7. doi: 10.1111/j.1754-9485.2011.02327.x. PMID 22339744
- [Background] Ambrosini V, Campana D, Tomassetti P, Grassetto G, Rubello D, Fanti S. PET/CT with 68Gallium-DOTA-peptides in NET: an overview. Eur J Radiol. 2011 Nov;80(2):e116-9. doi: 10.1016/j.ejrad.2010.07.022. Epub 2010 Aug 25. PMID 20800401
- [Background] Garcia C, Gebhart G, Flamen P. New PET imaging agents in the management of solid cancers. Curr Opin Oncol. 2012 Nov;24(6):748-55. doi: 10.1097/CCO.0b013e32835766f7. PMID 22913970
- [Background] Eisenhauer EA, Therasse P, Bogaerts J, Schwartz LH, Sargent D, Ford R, Dancey J, Arbuck S, Gwyther S, Mooney M, Rubinstein L, Shankar L, Dodd L, Kaplan R, Lacombe D, Verweij J. New response evaluation criteria in solid tumours: revised RECIST guideline (version 1.1). Eur J Cancer. 2009 Jan;45(2):228-47. doi: 10.1016/j.ejca.2008.10.026. PMID 19097774
- [Background] Sowa-Staszczak A, Chrzan R, Pach D, Stefanska A, Tomaszuk M, Buziak-Bereza M, Kolodziej M, Przybylik-Mazurek E, Hubalewska-Dydejczyk A. Are RECIST criteria sufficient to assess response to therapy in neuroendocrine tumors? Clin Imaging. 2012 Jul-Aug;36(4):360-4. doi: 10.1016/j.clinimag.2011.11.005. Epub 2012 Jun 8. PMID 22726975
- [Background] Panagiotidis E, Alshammari A, Michopoulou S, Skoura E, Naik K, Maragkoudakis E, Mohmaduvesh M, Al-Harbi M, Belda M, Caplin ME, Toumpanakis C, Bomanji J. Comparison of the Impact of 68Ga-DOTATATE and 18F-FDG PET/CT on Clinical Management in Patients with Neuroendocrine Tumors. J Nucl Med. 2017 Jan;58(1):91-96. doi: 10.2967/jnumed.116.178095. Epub 2016 Aug 11. PMID 27516446
- [Background] Johnbeck CB, Knigge U, Langer SW, Loft A, Berthelsen AK, Federspiel B, Binderup T, Kjaer A. Prognostic Value of 18F-FLT PET in Patients with Neuroendocrine Neoplasms: A Prospective Head-to-Head Comparison with 18F-FDG PET and Ki-67 in 100 Patients. J Nucl Med. 2016 Dec;57(12):1851-1857. doi: 10.2967/jnumed.116.174714. Epub 2016 Jul 28. PMID 27469355
- [Background] Abdulrezzak U, Kurt YK, Kula M, Tutus A. Combined imaging with 68Ga-DOTA-TATE and 18F-FDG PET/CT on the basis of volumetric parameters in neuroendocrine tumors. Nucl Med Commun. 2016 Aug;37(8):874-81. doi: 10.1097/MNM.0000000000000522. PMID 27096719
- [Background] Severi S, Nanni O, Bodei L, Sansovini M, Ianniello A, Nicoletti S, Scarpi E, Matteucci F, Gilardi L, Paganelli G. Role of 18FDG PET/CT in patients treated with 177Lu-DOTATATE for advanced differentiated neuroendocrine tumours. Eur J Nucl Med Mol Imaging. 2013 Jun;40(6):881-8. doi: 10.1007/s00259-013-2369-z. Epub 2013 Feb 27. PMID 23443937
- [Background] Valkema R, De Jong M, Bakker WH, Breeman WA, Kooij PP, Lugtenburg PJ, De Jong FH, Christiansen A, Kam BL, De Herder WW, Stridsberg M, Lindemans J, Ensing G, Krenning EP. Phase I study of peptide receptor radionuclide therapy with [In-DTPA]octreotide: the Rotterdam experience. Semin Nucl Med. 2002 Apr;32(2):110-22. doi: 10.1053/snuc/2002.31025. PMID 11965606
- [Background] Baur B, Solbach C, Andreolli E, Winter G, Machulla HJ, Reske SN. Synthesis, Radiolabelling and In Vitro Characterization of the Gallium-68-, Yttrium-90- and Lutetium-177-Labelled PSMA Ligand, CHX-A''-DTPA-DUPA-Pep. Pharmaceuticals (Basel). 2014 Apr 29;7(5):517-29. doi: 10.3390/ph7050517. PMID 24787458
- [Background] Otte A, Herrmann R, Heppeler A, Behe M, Jermann E, Powell P, Maecke HR, Muller J. Yttrium-90 DOTATOC: first clinical results. Eur J Nucl Med. 1999 Nov;26(11):1439-47. PMID 10552085
- [Background] Otte A, Mueller-Brand J, Dellas S, Nitzsche EU, Herrmann R, Maecke HR. Yttrium-90-labelled somatostatin-analogue for cancer treatment. Lancet. 1998 Feb 7;351(9100):417-8. doi: 10.1016/s0140-6736(05)78355-0. No abstract available. PMID 9482300
- [Background] Waldherr C, Pless M, Maecke HR, Haldemann A, Mueller-Brand J. The clinical value of [90Y-DOTA]-D-Phe1-Tyr3-octreotide (90Y-DOTATOC) in the treatment of neuroendocrine tumours: a clinical phase II study. Ann Oncol. 2001 Jul;12(7):941-5. doi: 10.1023/a:1011160913619. PMID 11521799
- [Background] Waldherr C, Pless M, Maecke HR, Schumacher T, Crazzolara A, Nitzsche EU, Haldemann A, Mueller-Brand J. Tumor response and clinical benefit in neuroendocrine tumors after 7.4 GBq (90)Y-DOTATOC. J Nucl Med. 2002 May;43(5):610-6. PMID 11994522
- [Background] Chinol M, Bodei L, Cremonesi M, Paganelli G. Receptor-mediated radiotherapy with Y-DOTA-DPhe-Tyr-octreotide: the experience of the European Institute of Oncology Group. Semin Nucl Med. 2002 Apr;32(2):141-7. doi: 10.1053/snuc.2002.31563. PMID 11965609
- [Background] Valkema R, Pauwels S, Kvols LK, Barone R, Jamar F, Bakker WH, Kwekkeboom DJ, Bouterfa H, Krenning EP. Survival and response after peptide receptor radionuclide therapy with [90Y-DOTA0,Tyr3]octreotide in patients with advanced gastroenteropancreatic neuroendocrine tumors. Semin Nucl Med. 2006 Apr;36(2):147-56. doi: 10.1053/j.semnuclmed.2006.01.001. PMID 16517236
- [Background] van der Zwan WA, Bodei L, Mueller-Brand J, de Herder WW, Kvols LK, Kwekkeboom DJ. GEPNETs update: Radionuclide therapy in neuroendocrine tumors. Eur J Endocrinol. 2015 Jan;172(1):R1-8. doi: 10.1530/EJE-14-0488. Epub 2014 Aug 12. PMID 25117465
- [Background] Paganelli G, Bodei L, Handkiewicz Junak D, Rocca P, Papi S, Lopera Sierra M, Gatti M, Chinol M, Bartolomei M, Fiorenza M, Grana C. 90Y-DOTA-D-Phe1-Try3-octreotide in therapy of neuroendocrine malignancies. Biopolymers. 2002;66(6):393-8. doi: 10.1002/bip.10349. PMID 12658726
- [Background] Bodei L, Cremonesi M, Zoboli S, Grana C, Bartolomei M, Rocca P, Caracciolo M, Macke HR, Chinol M, Paganelli G. Receptor-mediated radionuclide therapy with 90Y-DOTATOC in association with amino acid infusion: a phase I study. Eur J Nucl Med Mol Imaging. 2003 Feb;30(2):207-16. doi: 10.1007/s00259-002-1023-y. Epub 2002 Nov 16. PMID 12552338
- [Background] Valkema R, Pauwels SA, Kvols LK, Kwekkeboom DJ, Jamar F, de Jong M, Barone R, Walrand S, Kooij PP, Bakker WH, Lasher J, Krenning EP. Long-term follow-up of renal function after peptide receptor radiation therapy with (90)Y-DOTA(0),Tyr(3)-octreotide and (177)Lu-DOTA(0), Tyr(3)-octreotate. J Nucl Med. 2005 Jan;46 Suppl 1:83S-91S. PMID 15653656
- [Background] Imhof A, Brunner P, Marincek N, Briel M, Schindler C, Rasch H, Macke HR, Rochlitz C, Muller-Brand J, Walter MA. Response, survival, and long-term toxicity after therapy with the radiolabeled somatostatin analogue [90Y-DOTA]-TOC in metastasized neuroendocrine cancers. J Clin Oncol. 2011 Jun 10;29(17):2416-23. doi: 10.1200/JCO.2010.33.7873. Epub 2011 May 9. PMID 21555692
- [Background] Bodei L, Cremonesi M, Ferrari M, Pacifici M, Grana CM, Bartolomei M, Baio SM, Sansovini M, Paganelli G. Long-term evaluation of renal toxicity after peptide receptor radionuclide therapy with 90Y-DOTATOC and 177Lu-DOTATATE: the role of associated risk factors. Eur J Nucl Med Mol Imaging. 2008 Oct;35(10):1847-56. doi: 10.1007/s00259-008-0778-1. Epub 2008 Apr 22. PMID 18427807
- [Background] Guerriero F, Ferrari ME, Botta F, Fioroni F, Grassi E, Versari A, Sarnelli A, Pacilio M, Amato E, Strigari L, Bodei L, Paganelli G, Iori M, Pedroli G, Cremonesi M. Kidney dosimetry in (1)(7)(7)Lu and (9)(0)Y peptide receptor radionuclide therapy: influence of image timing, time-activity integration method, and risk factors. Biomed Res Int. 2013;2013:935351. doi: 10.1155/2013/935351. Epub 2013 Jun 20. PMID 23865075
- [Background] Cremonesi M, Ferrari M, Di Dia A, Botta F, De Cicco C, Bodei L, Paganelli G. Recent issues on dosimetry and radiobiology for peptide receptor radionuclide therapy. Q J Nucl Med Mol Imaging. 2011 Apr;55(2):155-67. PMID 21386788
- [Background] Kwekkeboom DJ, de Herder WW, Kam BL, van Eijck CH, van Essen M, Kooij PP, Feelders RA, van Aken MO, Krenning EP. Treatment with the radiolabeled somatostatin analog [177 Lu-DOTA 0,Tyr3]octreotate: toxicity, efficacy, and survival. J Clin Oncol. 2008 May 1;26(13):2124-30. doi: 10.1200/JCO.2007.15.2553. PMID 18445841
- [Background] Kwekkeboom DJ, Kam BL, van Essen M, Teunissen JJ, van Eijck CH, Valkema R, de Jong M, de Herder WW, Krenning EP. Somatostatin-receptor-based imaging and therapy of gastroenteropancreatic neuroendocrine tumors. Endocr Relat Cancer. 2010 Jan 29;17(1):R53-73. doi: 10.1677/ERC-09-0078. Print 2010 Mar. PMID 19995807
- [Background] Ezziddin S, Khalaf F, Vanezi M, Haslerud T, Mayer K, Al Zreiqat A, Willinek W, Biersack HJ, Sabet A. Outcome of peptide receptor radionuclide therapy with 177Lu-octreotate in advanced grade 1/2 pancreatic neuroendocrine tumours. Eur J Nucl Med Mol Imaging. 2014 May;41(5):925-33. doi: 10.1007/s00259-013-2677-3. Epub 2014 Feb 7. PMID 24504504
- [Background] NETTER-1 Phase III in Patients With Midgut Neuroendocrine Tumors Treated With 177Lu-DOTATATE: Efficacy and Safety Results. Clin Adv Hematol Oncol. 2016 May;14(5 Suppl 7):8-9. No abstract available. PMID 27168104
- [Background] Strosberg J, El-Haddad G, Wolin E, Hendifar A, Yao J, Chasen B, Mittra E, Kunz PL, Kulke MH, Jacene H, Bushnell D, O'Dorisio TM, Baum RP, Kulkarni HR, Caplin M, Lebtahi R, Hobday T, Delpassand E, Van Cutsem E, Benson A, Srirajaskanthan R, Pavel M, Mora J, Berlin J, Grande E, Reed N, Seregni E, Oberg K, Lopera Sierra M, Santoro P, Thevenet T, Erion JL, Ruszniewski P, Kwekkeboom D, Krenning E; NETTER-1 Trial Investigators. Phase 3 Trial of 177Lu-Dotatate for Midgut Neuroendocrine Tumors. N Engl J Med. 2017 Jan 12;376(2):125-135. doi: 10.1056/NEJMoa1607427. PMID 28076709
- [Background] Teunissen JJ, Kwekkeboom DJ, de Jong M, Esser JP, Valkema R, Krenning EP. Endocrine tumours of the gastrointestinal tract. Peptide receptor radionuclide therapy. Best Pract Res Clin Gastroenterol. 2005 Aug;19(4):595-616. doi: 10.1016/j.bpg.2005.04.001. PMID 16183530
- [Background] de Jong M, Breeman WA, Valkema R, Bernard BF, Krenning EP. Combination radionuclide therapy using 177Lu- and 90Y-labeled somatostatin analogs. J Nucl Med. 2005 Jan;46 Suppl 1:13S-7S. PMID 15653647
- [Background] Kunikowska J, Krolicki L, Hubalewska-Dydejczyk A, Mikolajczak R, Sowa-Staszczak A, Pawlak D. Clinical results of radionuclide therapy of neuroendocrine tumours with 90Y-DOTATATE and tandem 90Y/177Lu-DOTATATE: which is a better therapy option? Eur J Nucl Med Mol Imaging. 2011 Oct;38(10):1788-97. doi: 10.1007/s00259-011-1833-x. Epub 2011 May 7. PMID 21553086
- [Background] Seregni E, Maccauro M, Chiesa C, Mariani L, Pascali C, Mazzaferro V, De Braud F, Buzzoni R, Milione M, Lorenzoni A, Bogni A, Coliva A, Lo Vullo S, Bombardieri E. Treatment with tandem [90Y]DOTA-TATE and [177Lu]DOTA-TATE of neuroendocrine tumours refractory to conventional therapy. Eur J Nucl Med Mol Imaging. 2014 Feb;41(2):223-30. doi: 10.1007/s00259-013-2578-5. PMID 24233003
- [Background] Romer A, Seiler D, Marincek N, Brunner P, Koller MT, Ng QK, Maecke HR, Muller-Brand J, Rochlitz C, Briel M, Schindler C, Walter MA. Somatostatin-based radiopeptide therapy with [177Lu-DOTA]-TOC versus [90Y-DOTA]-TOC in neuroendocrine tumours. Eur J Nucl Med Mol Imaging. 2014 Feb;41(2):214-22. doi: 10.1007/s00259-013-2559-8. Epub 2013 Oct 2. PMID 24085501
- [Background] Bodei L, Cremonesi M, Grana CM, Chinol M, Baio SM, Severi S, Paganelli G. Yttrium-labelled peptides for therapy of NET. Eur J Nucl Med Mol Imaging. 2012 Feb;39 Suppl 1:S93-102. doi: 10.1007/s00259-011-2002-y. PMID 22388625
- [Background] Bodei L, Cremonesi M, Paganelli G. Yttrium-based therapy for neuroendocrine tumors. PET Clin. 2014 Jan;9(1):71-82. doi: 10.1016/j.cpet.2013.10.001. PMID 25029936
- [Background] Nisa L, Savelli G, Giubbini R. Yttrium-90 DOTATOC therapy in GEP-NET and other SST2 expressing tumors: a selected review. Ann Nucl Med. 2011 Feb;25(2):75-85. doi: 10.1007/s12149-010-0444-0. Epub 2010 Nov 25. PMID 21107762
- [Background] de Keizer B, van Aken MO, Feelders RA, de Herder WW, Kam BL, van Essen M, Krenning EP, Kwekkeboom DJ. Hormonal crises following receptor radionuclide therapy with the radiolabeled somatostatin analogue [177Lu-DOTA0,Tyr3]octreotate. Eur J Nucl Med Mol Imaging. 2008 Apr;35(4):749-55. doi: 10.1007/s00259-007-0691-z. Epub 2008 Jan 16. PMID 18210106
- [Background] Teunissen JJ, Kwekkeboom DJ, Kooij PP, Bakker WH, Krenning EP. Peptide receptor radionuclide therapy for non-radioiodine-avid differentiated thyroid carcinoma. J Nucl Med. 2005 Jan;46 Suppl 1:107S-14S. PMID 15653659
- [Background] Kwekkeboom DJ, Mueller-Brand J, Paganelli G, Anthony LB, Pauwels S, Kvols LK, O'dorisio TM, Valkema R, Bodei L, Chinol M, Maecke HR, Krenning EP. Overview of results of peptide receptor radionuclide therapy with 3 radiolabeled somatostatin analogs. J Nucl Med. 2005 Jan;46 Suppl 1:62S-6S. PMID 15653653
- [Background] Maecke HR, Reubi JC. Somatostatin receptors as targets for nuclear medicine imaging and radionuclide treatment. J Nucl Med. 2011 Jun;52(6):841-4. doi: 10.2967/jnumed.110.084236. Epub 2011 May 13. PMID 21571797
- [Background] Sun W, Lipsitz S, Catalano P, Mailliard JA, Haller DG; Eastern Cooperative Oncology Group. Phase II/III study of doxorubicin with fluorouracil compared with streptozocin with fluorouracil or dacarbazine in the treatment of advanced carcinoid tumors: Eastern Cooperative Oncology Group Study E1281. J Clin Oncol. 2005 Aug 1;23(22):4897-904. doi: 10.1200/JCO.2005.03.616. PMID 16051944
- [Background] Kouvaraki MA, Ajani JA, Hoff P, Wolff R, Evans DB, Lozano R, Yao JC. Fluorouracil, doxorubicin, and streptozocin in the treatment of patients with locally advanced and metastatic pancreatic endocrine carcinomas. J Clin Oncol. 2004 Dec 1;22(23):4762-71. doi: 10.1200/JCO.2004.04.024. PMID 15570077
- [Background] Raymond E, Dahan L, Raoul JL, Bang YJ, Borbath I, Lombard-Bohas C, Valle J, Metrakos P, Smith D, Vinik A, Chen JS, Horsch D, Hammel P, Wiedenmann B, Van Cutsem E, Patyna S, Lu DR, Blanckmeister C, Chao R, Ruszniewski P. Sunitinib malate for the treatment of pancreatic neuroendocrine tumors. N Engl J Med. 2011 Feb 10;364(6):501-13. doi: 10.1056/NEJMoa1003825. PMID 21306237
- [Background] Yao JC, Shah MH, Ito T, Bohas CL, Wolin EM, Van Cutsem E, Hobday TJ, Okusaka T, Capdevila J, de Vries EG, Tomassetti P, Pavel ME, Hoosen S, Haas T, Lincy J, Lebwohl D, Oberg K; RAD001 in Advanced Neuroendocrine Tumors, Third Trial (RADIANT-3) Study Group. Everolimus for advanced pancreatic neuroendocrine tumors. N Engl J Med. 2011 Feb 10;364(6):514-23. doi: 10.1056/NEJMoa1009290. PMID 21306238
- [Background] Baum RP, Kluge AW, Kulkarni H, Schorr-Neufing U, Niepsch K, Bitterlich N, van Echteld CJ. [(177)Lu-DOTA](0)-D-Phe(1)-Tyr(3)-Octreotide ((177)Lu-DOTATOC) For Peptide Receptor Radiotherapy in Patients with Advanced Neuroendocrine Tumours: A Phase-II Study. Theranostics. 2016 Feb 13;6(4):501-10. doi: 10.7150/thno.13702. eCollection 2016. PMID 26941843
- [Background] Schuchardt C, Kulkarni HR, Prasad V, Zachert C, Muller D, Baum RP. The Bad Berka dose protocol: comparative results of dosimetry in peptide receptor radionuclide therapy using (177)Lu-DOTATATE, (177)Lu-DOTANOC, and (177)Lu-DOTATOC. Recent Results Cancer Res. 2013;194:519-36. doi: 10.1007/978-3-642-27994-2_30. PMID 22918780
- [Background] Kratochwil C, Lopez-Benitez R, Mier W, Haufe S, Isermann B, Kauczor HU, Choyke PL, Haberkorn U, Giesel FL. Hepatic arterial infusion enhances DOTATOC radiopeptide therapy in patients with neuroendocrine liver metastases. Endocr Relat Cancer. 2011 Sep 20;18(5):595-602. doi: 10.1530/ERC-11-0144. Print 2011 Oct. PMID 21791571
- [Background] Paganelli G, Zoboli S, Cremonesi M, Bodei L, Ferrari M, Grana C, Bartolomei M, Orsi F, De Cicco C, Macke HR, Chinol M, de Braud F. Receptor-mediated radiotherapy with 90Y-DOTA-D-Phe1-Tyr3-octreotide. Eur J Nucl Med. 2001 Apr;28(4):426-34. doi: 10.1007/s002590100490. PMID 11357492